CLINICAL TRIAL: NCT03447366
Title: Assessment of Mitral Doppler as a Predictor of Respiratory Worsening After Vascular Filling for ICU Patients With Mechanical Ventilation. The EVALDM Study
Brief Title: Mitral Doppler as a Predictor of Respiratory Worsening After Vascular Filling
Acronym: EVALDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHMS17002
Record Dates: First submitted 2018-02-02; First posted 2018-02-27 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Respiration, Artificial; Vascular Filling; Echocardiography
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitral doppler (Experimental): Mitral doppler before and after vascular filling
  Interventions: Diagnostic Test: mitral doppler

INTERVENTIONS:
Diagnostic Test: mitral doppler — Mitral doppler before and after vascular filling

SUMMARY:
Interventional study of the accuracy of a non-invasive testing by echocardiography to predict respiratory worsening after vascular filling.

DETAILED DESCRIPTION:
Mitral Doppler will be performed before vascular filling. Patients will be classified in two groups (normal or high cardiac filling pressure).

The evolution of the respiratory data (SpO2/FiO2) of the two groups of the patients before and after vascular filling will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation
* And hemodynamic failure
* And decision of the attending physician to perform a vascular filling

Exclusion Criteria:

* Pregnancy and breast-feeding women
* Patients deprived of their administrative or judicial freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
frequency of the occuring of premature degradation respiratory | 30 minutes after vascular filling
  definied by a reduction of at least 15% of the SpO2/FiO2 ratio in the 30min following the vascular filling

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Ch Bourg En Bresse, Bourg-en-Bresse
  - Centre Hospitalier Metropole Savoie, Chambéry
  - CHU Grenoble Alpes, La Tronche

IPD SHARING:
Plan to Share IPD: No